CLINICAL TRIAL: NCT05092737
Title: Physiological Response to Prone Position in Intubated Adults With COVID-19 Associated Acute Respiratory Distress Syndrome (ARDS): a Retrospective Study
Brief Title: Physiological Response to Prone Position in COVID-19 Associated Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Piquilloud Imboden Lise, Principal Investigator, University of Lausanne Hospitals
Other Study IDs: Prone_COVID
Record Dates: First submitted 2021-10-21; First posted 2021-10-25 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2021-10

CONDITIONS: ARDS; Sars-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Prone positioning — Prone position during invasive mechanical ventilation

SUMMARY:
Retrospective study in COVID-19 ARDS patients hospitalised in the ICU. Investigators aim to explore the effects of prone positioning on oxygenation, dead space ventilation and mortality.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 associated moderate to severe ARDS
* Invasive mechanical ventilation
* Prone positioning
* admitted to ICU

Exclusion Criteria:

* already sustained prone positioning in referring hospital
* pronation during ECMO only
* denied consent for data analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 moderate to severe ARDS patients who sustained prone positioning
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 | Within 2 hours before pronation and 2 hours before supination
  Arterial partial pressure of oxygen / Fraction of inspired oxygen

SECONDARY OUTCOMES:
Alveolo-arterial oxygen gradient change | Within 2 hours before pronation and 2 hours before supination
Ventilatory Ratio | Within 2 hours before pronation and 2 hours before supination
Mortality or Extracorporeal membrane oxygenation (ECMO) support | Once between ICU admission and extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Lausanne University Hospitals, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No